CLINICAL TRIAL: NCT06537635
Title: The Impact of a Seated Compact Elliptical on Vital Signs and Range of Motion During Thirty Minutes of Activity
Brief Title: Cubii Vital Sign and Range of Motion Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CubiiPro
Record Dates: First submitted 2023-04-18; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Effects of; Exertion
Keywords: compact elliptical; range of motion; aerobic exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 30-minute session of exercise using a seated compact elliptical trainer (Experimental)
  Interventions: Device: Cubii seated compact elliptical trainer

INTERVENTIONS:
Device: Cubii seated compact elliptical trainer — The Cubii® Pro is an under-desk seated elliptical trainer. This device provides 8 levels of resistance and documents the total number of strides, distance covered in miles, and calories expended during an activity session.

SUMMARY:
The purpose of this study is to evaluate the effect of a seated compact elliptical on vital signs and range of motion (of knees and ankles) following thirty minutes of activity.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of 30 minutes of exercise on a seated compact elliptical on vital signs and range of motion (ROM). A convenience sample of 40 patients will be recruited for this study in two phases. The first phase from younger 18-30 staff from Kaizo Health who currently engage in a program or aerobic exercise greater than 90 minutes per week and report no previously diagnosed chronic health problems. Phase two will take place among the patient population of Kaizo Health consisting of men and women between 30-70. The purpose of recruiting in two phases is generate a more diverse sample. Participants must be able to perform all study procedures in order to participate. Exclusionary criteria will include less than 18 years of age, pregnancy, cancer, or the any of the conditions on the ACSM absolute and relative contraindications to exercise. After explanation of the study and consent is obtained, participants will complete the demographics form, medication questionnaire, the Self-Administered Comorbidity Questionnaire, and International Physical Activity Questionnaire short form. After completing the initial paperwork, participant's vital signs (blood pressure, heart rate, and oxygen saturation) and ROM of the ankle and knee will be assessed (T1). Following baseline measures, participants will perform a one-minute warm-up, thirty minutes of activity, and a two-minute cool-down on the Cubii®, a seated compact elliptical. During all activity, heart rate and oxygen saturation will be recorded every minute. Following the cooldown, blood pressure, heart rate, oxygen saturation, and ROM will be reassessed (T2). At the end of T2, steps, elliptical strides, distance, time, and calories burned will be recorded from the Cubii®. Additionally, all participants will complete a satisfaction questionnaire about the Cubii®.

ELIGIBILITY:
Inclusion Criteria:

* currently engage in a program or aerobic exercise greater than 90 minutes per week
* report no previously diagnosed chronic health problems
* patient population of Kaizo Health
* perform all study procedures in order to participate

Exclusion Criteria:

* less than 18 years of age
* pregnancy
* cancer
* any of the conditions on the ACSM absolute and relative contraindications to exercise

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Overall Satisfaction | After the 30-minute treatment (T4)
  The Customer Satisfaction (CSAT) was measured to gain insights into the patients' satisfaction of using the Cubii®. This CSAT asks a series of questions related to the ease of use, comfort, side effects, and overall satisfaction of the device. The participant responds by rating each question on a scale of 1 to 5, 1 being very unsatisfied, 2 being unsatisfied, 3 being neutral, 4 satisfied, and 5 very satisfied.
Ease of Use | After the 30-minute treatment (T4)
  The Customer Satisfaction (CSAT) was measured to gain insights into the patients' satisfaction of using the Cubii®. This CSAT asks a series of questions related to the ease of use, comfort, side effects, and overall satisfaction of the device. The participant responds by rating each question on a scale of 1 to 5, 1 being very unsatisfied, 2 being unsatisfied, 3 being neutral, 4 satisfied, and 5 very satisfied.
Refer a friend | After the 30-minute treatment (T4)
  The Customer Satisfaction (CSAT) was measured to gain insights into the patients' satisfaction of using the Cubii®. This CSAT asks a series of questions related to the ease of use, comfort, side effects, and overall satisfaction of the device. The participant responds by rating each question on a scale of 1 to 5, 1 being very unsatisfied, 2 being unsatisfied, 3 being neutral, 4 satisfied, and 5 very satisfied.
Knee Flexion Baseline | This information was collected after the 30-minute treatment (T4).
  Knee flexion range of motion was evaluated using the EasyAngle, a digital goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Spine Rehab, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No